CLINICAL TRIAL: NCT03734913
Title: A Phase 1, Open-Label, Dose-Escalation and Expansion, Safety and Tolerability Study of ZSP1602 in Participants With Advanced Solid Tumors
Brief Title: A Phase 1 Study of ZSP1602 in Participants With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Zhongsheng Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZSP1602-16-01
Record Dates: First submitted 2018-11-05; First posted 2018-11-08 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Basal Cell Carcinoma; Medulloblastoma; Adenocarcinoma of Esophagogastric Junction; Small Cell Lung Cancer; Neuroendocrine Neoplasm; Glioblastoma
MeSH Terms: conditions — Carcinoma, Basal Cell; Medulloblastoma; Small Cell Lung Carcinoma; Neuroendocrine Tumors; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): Participants with advanced solid tumors including basal cell carcinoma and medulloblastoma, regardless of SMO or Gli1 alteration status.
  Interventions: Drug: ZSP1602
- Part 2 Cohort A (Experimental): Participants with Adenocarcinoma of Esophagogastric Junction with SMO or Gli1 protein overexpression alteration.
  Interventions: Drug: ZSP1602
- Part 2 Cohort B (Experimental): Participants with basal cell carcinoma, small cell lung cancer, neuroendocrine neoplasm and glioblastoma with SMO or Gli1 protein overexpression alteration.
  Interventions: Drug: ZSP1602

INTERVENTIONS:
Drug: ZSP1602 — ZSP1602 capsules for oral administration

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics, and determine the maximum tolerated dose of ZSP1602 in participants with basal cell carcinoma, adenocarcinoma of esophagogastric junction, small cell lung cancer, neuroendocrine neoplasm and other advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants are required to meet all the criteria below in order to be included in the trial:

  1. Male or female participants, aged 18 ~ 75 years.

     Confirmed diagnosis of advanced solid tumors by histological or cytological examination, Participants have no effective standard anticancer therapy available or is intolerant to standard anticancer therapy. For Part 1 Dose Ascending Stage, and Part 2 Dose expansion Stage:

     For Part 1: Advanced solid tumors including basal cell carcinoma and medulloblastoma, regardless of SMO or Gli1 alteration status.

     For Part 2: Participants will be enrolled into cohort A and cohort B. Cohort A: Participants with Adenocarcinoma of Esophagogastric Junction with SMO or Gli1 protein overexpression alteration. (IHC≥1%) Cohort B: Participants with basal cell carcinoma, small cell lung cancer, neuroendocrine neoplasm and glioblastoma with SMO or Gli1 protein overexpression alteration. (IHC≥1%)
  2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
  3. Participants with at least 1 measurable tumor lesion based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1) and response assessment in neuro-oncology criteria (RANO) (participants with glioblastoma must accept skull MRI scanning.)
  4. Recovery from past medical history of adverse reactions (excluding alopecia and neurotoxicity) caused by radiotherapy and chemotherapy to national cancer institute common terminology criteria for adverse events 4.03 (NCI CTCAE 4.03) ≤Grade 1 or baseline level.
  5. Life expectancy > 12 weeks.
  6. Adequate organ function, defined by the following laboratory results, to be obtained prior to registration and enrollment:

     Bone marrow function: absolute neutrophil count (ANC)≥1.5×10^9/L; hemoglobin (HB)≥90 g/L; Platelet count (PLT)≥75×10^9/L.

     Liver function: Alanine aminotransferase (ALT)≤2.5×the upper limit of normal (ULN), aspartate aminotransferase (AST)≤2.5×ULN, alkaline phosphatase (ALP)≤2.5×ULN, total bilirubin (TBIL)≤1.5×ULN; ALT≤5×ULN, AST≤5×ULN, ALP≤5×ULN (For participants with liver metastasis).

     Renal function: creatinine≤1.5×ULN; clearance (CL)≥ 60 mL/min. Coagulation function: international normalized ratio (INR)≤1.5×ULN, activated partial thromboplastin time (APTT)≤1.5×ULN.

     Left ventricular ejection fractions (LVEF)≥50%. Creatine kinase (CK)≤2.5×ULN.
  7. Participants (including partners) have no gestation plans and must use reliable methods of contraception during the study and until 8 months following the last dose of investigational product.
  8. Participants must provide a written dated Informed Consent Form (ICF) with signature prior to screening.
  9. Participants must be willing and able to adhere to the visit schedule and protocol requirements and be available to complete the study.

Exclusion Criteria:

* Eligible participants must not meet any of the following exclusion criteria:

  1. Participants who have intracranial tumor and/or brain metastases with clinical symptoms and need treatment are ineligible except for the following circumstances:

     1. recovery from the therapy (including radiotherapy and/or surgery) 4 weeks before enrollment.
     2. Participants with intracranial tumor who are clinically stable during screening and enrollment, have no need to medication by hormone or anticonvulsants, and are estimated to be clinically stable during the study.
  2. Participants with glioblastoma confirmed diagnosis via MRI or CT of intracranial hemorrhage and intratumor hemorrhage.
  3. Participants with positive human immunodeficiency virus(HIV) or hepatitis C virus antibody (HCV) or hepatitis B surface antigen (HBV DNA>2.0 ×103 IU/ml) or active infections which require systematic antibiotics therapy or concurred with unexplainable fever before drug treatment.
  4. History of pulmonary fibrosis or interstitial pneumonia including pneumoconiosis and radiation pulmonary fibrosis beyond radiation field.
  5. Participants with dysphagia.
  6. Participants with incontrollable hydrops in third lumen such as malignant pleural effusion and ascites.
  7. Participants with Diarrhea > Grade 2 (according to CTCAE 4.03)
  8. Any clinically significant gastrointestinal abnormalities, which may impair absorption of ZSP1602, such as Crohn's disease, ulcerative colitis and subtotal gastrectomy.
  9. Participants with major surgery or active peptic ulcer disease or unrecovered wound.
  10. History of myocardial infarction or congestive heart-failure (CHF) at NYHA≥3 level within 6 months prior to enrollment.
  11. Has either a history of uncontrollable or unstable angina pectoris or a history of severe or uncontrollable ventricular arrhythmia.
  12. Participants with QTcF prolongations in electrocardiogram (ECG) baseline (QTcF>450ms for males or QTcF>470ms for females) or with high risk factors leading to QT intervals prolonging (including hypokalemia, familial QT interval prolongation syndrome).
  13. Participants with concomitant illness such as hemorrhagic or thrombotic diseases or with anticoagulant treatment in routine dose for the moment.
  14. Participants with medications known to be moderate and strong inhibitors or inducers of CYP3A4 during screening and that cannot be discontinued before starting treatment with ZSP1602.
  15. History of most recently chemotherapy, radiotherapy, or non-antibody antitumor biologics within 4 weeks prior to the first ZSP1602 treatment and last time medication of nitrosoureas, mitomycin C or doxorubicin within 6 weeks and latest usage of antibody antitumor biologics within 8 weeks.
  16. History of autoimmune disease.
  17. History of allergic reactions to ZSP1602, any of the excipients of ZSP1602 or similar compounds.
  18. Pregnant or nursing women.
  19. Participants who, in the judgment of the investigator, will be unfit for the study. ( For reasons such as poor compliance, unsuitable for venous catheterization and so on)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2019-01-25 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity (DLT) | At day 32 after first dosing.
  To determine the DLT of ZSP1602 in advanced solid tumor participants accessed by CTCAE4.03
Maximum tolerated dose (MTD) | At day 32 after first dosing.
  The highest dose at the level with <= 2/6 participants experienced DLT.

SECONDARY OUTCOMES:
Time to progression (TTP) | From Screening, Day 28 of Cycle1 (28 days), then every 8 weeks, until disease progression or discontinuation from study (approximately 18 months or earlier if participants terminate from the study).
  For Part1 and Part2
Over all response (ORR) | From Screening, Day 28 of Cycle1 (28 days), then every 8 weeks, until disease progression or discontinuation from study (approximately 18 months or earlier if participants terminate from the study).
  For Part1 and Part2
Cmax of ZSP1602 | Protocol-defined time points during Cycles 0 (4 days) and 1 (28 days) of treatment per participants.
  For Part1 and Part2
Tmax of ZSP1602 | Protocol-defined time points during Cycles 0 (4 days) and 1 (28 days) of treatment per participants.
  For Part1 and Part2
Cmin of ZSP1602 | Protocol-defined time points during Cycles 0 (4 days) and 1 (28 days) of treatment per participants.
  For Part1 and Part2
AUC0-t of ZSP1602 | Protocol-defined time points during Cycles 0 (4 days) and 1 (28 days) of treatment per participants.
  For Part1 and Part2
T1/2 of ZSP1602 | Protocol-defined time points during Cycles 0 (4 days) and 1 (28 days) of treatment per participants.
  For Part1 and Part2
Cl/F of ZSP1602 | Protocol-defined time points during Cycles 0 (4 days) and 1 (28 days) of treatment per participants.
  For Part1 and Part2

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin Cancer Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No